CLINICAL TRIAL: NCT04211792
Title: Comparison of Intraocular Pressure Measurements Between Icare PRO, Icare ic200, and Goldmann Applanation Tonometer
Brief Title: IOP Device Comparison Study
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: Tonometry
Record Dates: First submitted 2019-12-21; First posted 2019-12-26 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2020-06

CONDITIONS: Intraocular Pressure
Keywords: Tonometry, Ocular; Concordance; Intraocular Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glaucoma suspect or patients: Patients who has or suspected Glaucoma will be approached for the recruitment into this study. IOP will be measured in the sitting position with Icare tonometers in a random order in both the eyes. IOP measurements by GAT will be taken after Icare measurements followed by CCT recording with ultrasound pachymeter.
  Interventions: Device: Icare Tonometer

INTERVENTIONS:
Device: Icare Tonometer — Icare tonometers are a new class of rebound tonometers for IOP measurements. The Icare series of tonometers are hand-held tonometers, which are easy to operate and generally do not require topical anaesthesia for IOP measurements.

SUMMARY:
Intraocular pressure measurement (IOP) is part of a routine eye examination. High and low eye pressure may be linked to certain eye conditions such as glaucoma. The current gold standard for IOP measurement is a technique called Goldmann Applanation Tonometry (GAT). GAT requires the use of a Goldmann applanation tonometer mounted on a slit lamp. Apart from GAT, there are many other devices that can be used to measure IOP, including the iCare tonometers. In this prospective study, investigators will be measuring participant's IOP with GAT, Icare PRO, and Icare ic200 tonometers to see if there is an agreement in IOP between the different devices. Investigator will also look if there is a concordance between different tonometers in low, moderate and high IOP range. Given the postural requirements for performing GAT, patients with higher body mass index (BMI) tend to have difficulties with proper positioning at the slit lamp that may lead to inaccurate GAT measurements. To this end, investigators will analyze the effect of BMI on IOP measurements with different devices. Additionally, comfort level of the patients with different tonometry devices will be recorded using a visual analog scale.

DETAILED DESCRIPTION:
Intraocular pressure measurement (IOP) is a vital part of the routine eye examination. High and low eye pressure may be associated with various ocular pathologies, including glaucoma. The current gold standard for IOP measurement is Goldmann Applanation Tonometry (GAT). To perform measurements with GAT, topical anaesthetic and fluorescein eye drops are applied to the eye. The Goldmann tonometer tip directly contacts the cornea and measures the intraocular pressure by the Imbert-Fick principle. IOP measurement is generally performed by a trained and experienced ophthalmologist or ophthalmic technician on patients in an upright position. There may be minor discomfort associated with the use of topical anaesthetic in this technique.

Icare tonometers are a new class of rebound tonometers used for IOP measurements. A disposable tip of the Icare tonometer is propelled towards the cornea and the deceleration of the tip is measured to calculate the IOP. The Icare series of devices are hand-held tonometers, which are easy to operate and do not require topical anaesthesia for IOP measurements.

Despite being the most reliable and clinically validated method to measure IOP, GAT has several limitations. First, it requires extensive training and experience to accurately measure IOP. Moreover, IOP measurement with GAT may be associated with minor discomfort due to the need for topical anaesthesia. Apart from that, GAT is not a portable device and the patient needs to be seated upright, making it difficult to perform in certain populations, such as pediatric, elderly and those with high BMI. Several hand-held tonometers are available, including the Icare series. These tonometers allow for quick, portable, and arguably easier IOP measurements. These tonometers do not require as rigorous training to use. However, there is an inconsistency in the data to verify if the IOP measurements by Icare is in concordance with GAT measurements. Recent Meta-analysis by Rödter and colleagues neither confirm nor deny the agreement between Icare and GAT tonometers.

The purpose of the current study is to prospectively evaluate and determine the relationship of the IOP measurements obtained by Icare PRO, Icare ic200, and GAT. The study will evaluate IOP measurements in different IOP ranges (low: 7-15mmHg, Moderate: 16- 22mmHg, High: 23-60 mmHg) as well as the effects of central corneal thickness and BMI on IOP measurements. Patient comfort during tonometry will be measured using a visual analogue scale. To date, this will be the first study in Canada to compare IOP measurements between Icare PRO, Icare ic200, and GAT in different IOP ranges. Additionally, as the Icare ic200 is a new device, this will be the first study to perform a comparative functional analysis of the Icare ic200 versus GAT.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Willingness to participate in all study procedures, along with signed written consent

Exclusion Criteria:

* Age younger than 18 years
* Participants with corneal defects (edema, scarring, cicatrix, opacity)
* Participants with epithelial lesions, prior refractive surgery and keratoplasty surgery
* Participants having corneal astigmatism ≥ 3D
* Participants who wear contact lenses
* Participants with proliferative diabetic retinopathy, Uveitis
* Participants who are unable to have IOP measured by Goldmann Tonometry
* Inability to provide informed consent
* Participants with proliferative diabetic retinopathy, Uveitis
* Participation in a clinical trial with investigational products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma suspects or patients who are older than 18 years are invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Concordance in IOP between GAT and Icare ic200 | It's a single visit study and it is anticipated that study procedures will increase the duration of the clinic visit by 20 minutes.
  Primary objective of this study is to compare overall Mean IOP between GAT and Icare ic200

SECONDARY OUTCOMES:
Concordance in IOP between GAT and Icare PRO | It's a single visit study and it is anticipated that study procedures will increase the duration of the clinic visit by 20 minutes.
  To compare the overall IOP measurements between GAT and Icare PRO.
Concordance among tonometers in low IOP range | It's a single visit study and it is anticipated that study procedures will increase the duration of the clinic visit by 20 minutes.
  To compare IOP measurements between GAT and Icare PRO/Icare ic200 in low IOP range (7-15 mmHg).
Concordance among tonometers in medium IOP range | It's a single visit study and it is anticipated that study procedures will increase the duration of the clinic visit by 20 minutes.
  To compare IOP measurements between GAT and Icare PRO/Icare ic200 in medium IOP range (16-22 mmHg).
Concordance among tonometers in high IOP range | It's a single visit study and it is anticipated that study procedures will increase the duration of the clinic visit by 20 minutes.
  To compare IOP measurements between GAT and Icare PRO/Icare ic200 in high IOP range (23-60 mmHg).
Proportion of Icare IOP measurements with GAT recordings | It's a single visit study and it is anticipated that study procedures will increase the duration of the clinic visit by 20 minutes.
  To determine the proportion of IOP measurements from Icare PRO and Icare ic200 that are within ±2 mmHg, ±3 mmHg and ±5 mmHg of the GAT measurements.
Corelation between GAT and Icare Tonometers | It's a single visit study and it is anticipated that study procedures will increase the duration of the clinic visit by 20 minutes.
  To find the correlation in the IOP measurement between GAT and Icare PRO and also between GAT and Icare ic200.
Corelation between central corneal thickness (CCT) and IOP | It's a single visit study and it is anticipated that study procedures will increase the duration of the clinic visit by 20 minutes.
  To evaluate the effect of central corneal thickness (CCT) on IOP measurement by GAT, Icare PRO and Icare ic200.
Effect of BMI on IOP | It's a single visit study and it is anticipated that study procedures will increase the duration of the clinic visit by 20 minutes.
  To evaluate the effects of BMI on IOP measurement by GAT, Icare PRO, Icare ic200.
Patient comfort during tonometry | It's a single visit study and it is anticipated that study procedures will increase the duration of the clinic visit by 20 minutes.
  To evaluate patient comfort during tonometry measurements with each device using a Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lin, MD, Principal Investigator — Ivey Eye Institute- St Joseph's hospital
Locations (1):
- Ivey Eye Institute at St Joseph hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nakakura S. Icare(R) rebound tonometers: review of their characteristics and ease of use. Clin Ophthalmol. 2018 Jul 12;12:1245-1253. doi: 10.2147/OPTH.S163092. eCollection 2018. PMID 30034218
- [Result] Kass MA. Standardizing the measurement of intraocular pressure for clinical research. Guidelines from the Eye Care Technology Forum. Ophthalmology. 1996 Jan;103(1):183-5. doi: 10.1016/s0161-6420(96)30741-0. No abstract available. PMID 8628552
- [Result] Pakrou N, Gray T, Mills R, Landers J, Craig J. Clinical comparison of the Icare tonometer and Goldmann applanation tonometry. J Glaucoma. 2008 Jan-Feb;17(1):43-7. doi: 10.1097/IJG.0b013e318133fb32. PMID 18303384
- [Result] Kim KN, Jeoung JW, Park KH, Yang MK, Kim DM. Comparison of the new rebound tonometer with Goldmann applanation tonometer in a clinical setting. Acta Ophthalmol. 2013 Aug;91(5):e392-6. doi: 10.1111/aos.12109. Epub 2013 Mar 25. PMID 23521889
- [Result] Yildiz A, Yasar T. Comparison of Goldmann applanation, non-contact, dynamic contour and tonopen tonometry measurements in healthy and glaucomatous eyes, and effect of central corneal thickness on the measurement results. Med Glas (Zenica). 2018 Aug 1;15(2):152-157. doi: 10.17392/960-18. PMID 30047543
- [Result] Poostchi A, Mitchell R, Nicholas S, Purdie G, Wells A. The iCare rebound tonometer: comparisons with Goldmann tonometry, and influence of central corneal thickness. Clin Exp Ophthalmol. 2009 Sep;37(7):687-91. doi: 10.1111/j.1442-9071.2009.02109.x. PMID 19788665
- [Result] Grewal DS, Stinnett SS, Folgar FA, Schneider EW, Vajzovic L, Asrani S, Freedman SF, Mruthyunjaya P, Hahn P. A Comparative Study of Rebound Tonometry With Tonopen and Goldmann Applanation Tonometry Following Vitreoretinal Surgery. Am J Ophthalmol. 2016 Jan;161:22-8.e1-8. doi: 10.1016/j.ajo.2015.09.022. Epub 2015 Sep 25. PMID 26408266
- [Result] Rateb M, Abdel-Radi M, Eldaly Z, Elmohamady MN, Noor El Din A. Comparison of IOP Measurement by Goldmann Applanation Tonometer, ICare Rebound Tonometer, and Tono-Pen in Keratoconus Patients after MyoRing Implantation. J Ophthalmol. 2019 May 9;2019:1964107. doi: 10.1155/2019/1964107. eCollection 2019. PMID 31210982
- [Result] Nakakura S, Mori E, Fujio Y, Fujisawa Y, Matsuya K, Kobayashi Y, Tabuchi H, Asaoka R, Kiuchi Y. Comparison of the Intraocular Pressure Measured Using the New Rebound Tonometer Icare ic100 and Icare TA01i or Goldmann Applanation Tonometer. J Glaucoma. 2019 Feb;28(2):172-177. doi: 10.1097/IJG.0000000000001138. PMID 30689609
- [Result] Munkwitz S, Elkarmouty A, Hoffmann EM, Pfeiffer N, Thieme H. Comparison of the iCare rebound tonometer and the Goldmann applanation tonometer over a wide IOP range. Graefes Arch Clin Exp Ophthalmol. 2008 Jun;246(6):875-9. doi: 10.1007/s00417-007-0758-3. Epub 2008 Jan 12. PMID 18196259
- [Result] Brusini P, Salvetat ML, Zeppieri M, Tosoni C, Parisi L. Comparison of ICare tonometer with Goldmann applanation tonometer in glaucoma patients. J Glaucoma. 2006 Jun;15(3):213-7. doi: 10.1097/01.ijg.0000212208.87523.66. PMID 16778643
- [Result] Rodter TH, Knippschild S, Baulig C, Krummenauer F. Meta-analysis of the concordance of Icare(R) PRO-based rebound and Goldmann applanation tonometry in glaucoma patients. Eur J Ophthalmol. 2020 Mar;30(2):245-252. doi: 10.1177/1120672119866067. Epub 2019 Aug 29. PMID 31466475
- [Result] Schweier C, Hanson JV, Funk J, Toteberg-Harms M. Repeatability of intraocular pressure measurements with Icare PRO rebound, Tono-Pen AVIA, and Goldmann tonometers in sitting and reclining positions. BMC Ophthalmol. 2013 Sep 5;13:44. doi: 10.1186/1471-2415-13-44. PMID 24006952